CLINICAL TRIAL: NCT06965036
Title: Fattori di Rischio ed Outcome Dell'Ictus Ischemico da Occlusione Tandem di Circolo Anteriore e Posteriore
Brief Title: Risk Factors and Outcomes of Ischemic Stroke Associated With Tandem or Isolated Cervical Artery Occlusion in Anterior and Posterior Circulation
Acronym: CERES-TANDEM
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Unità Sanitaria Locale della Romagna (Other)
Collaborators: Hospital Universitari Vall d'Hebron Research Institute (Other); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Michele Romoli, Principal Investigator, Azienda Unità Sanitaria Locale della Romagna
Other Study IDs: 0001765/2024
Record Dates: First submitted 2025-04-25; First posted 2025-05-11 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Acute Ischemic Stroke Related to Tandem Occlusion; Acute Ischemic Stroke Due to Isolated Cervical Artery Occlusion
Keywords: stroke; tandem occlusion; cervical artery occlusion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- emergent carotid (or cervical artery) stenting: An aggressive approach characterized by stenting the extracranial occluded vessel (independently from the retrograde or anterograde approach) during the process of mechanical thrombectomy (hyperacute stage).
- conservative management: Any management except from emergent carotid stenting (conservative management)

SUMMARY:
CERES-TANDEM is a multicenter study designed to improve the understanding of "tandem" ischemic stroke -those caused by two blockages in series, one in a neck artery and one in a brain artery-. Because tandem occlusion-related stroke tend to cause more severe brain injury and have been under-represented in major clinical trials, there is no clear consensus on which treatments work best. This study will help identify who is most at risk and which therapies lead to the best recovery.

OBJECTIVES:

Identify Risk Factors: Compare common stroke risk factors (e.g., high blood pressure, diabetes, high cholesterol, smoking) in patients with tandem occlusion versus those with single-site large vessel occlusions.

Compare Clinical Outcomes of Reperfusion: Evaluate whether acute reperfusion treatments-such as clot-dissolving drugs (thrombolysis), mechanical clot removal (thrombectomy), and emergent carotid stenting-lead to better 3-month functional outcome (assessed by the modified Rankin Scale, ranging 0 to 6, with good functional outcome identified with mRS score 0-2) compared to medical management alone in tandem occlusion and isolated cervical artery occlusion.

Assess Post Stent Therapy: Among patients who receive emergent stenting, determine whether different post-stenting regimens (antiplatelet agents, anticoagulants, or no additional therapy) affect functional outcomes, bleeding events, or stroke recurrence.

STUDY DESIGN:

Type: cohort study pooling data from prospective registries of cerebrovascular diseases at participating sites Setting: Stroke Unit, Cesena Hospital (PI MR), Interventional Neuroradiology, Vall d'Hebron Research Institute, Barcelona (PI FD), Radiology, Boston Medical Center (PI TN); and other participating stroke centers Time Frame: Patients treated between 2018 and 2024. Sample Size: Approximately 2800 cases overall

DATA COLLECTION:

Sources: Clinical records, imaging reports (CT perfusion, angiograms), lab results, hospital discharge summaries, and longitudinale stroke registry databases.

Data Safety: case information is anonymized using encrypted study IDs; only aggregate data will be reported.

Follow-Up: Standard-of-care follow-up visits at 3 months (minimum) and up to 12 months or until death. Outcomes include functional status (mRS), recurrence of stroke or TIA, symptomatic intracranial hemorrhage, major bleeding, and all-cause mortality

OUTCOMES AND ANALYSIS:

Primary Outcome: Functional outcome, identified by the mRS and tested between groups with ordinal shift between mRS categories (0-6).

Secondary Outcomes: functional status at 3 months (excellent outcome mRS 0-1, good outcome mRS 0-2) Additional outcomes: early neurological deterioration; symptomatic intracerebral hemorrhage and successful recanalization (defined as TICI 2b or higher).

PLANNED ANALYSIS (see Detailed Description for full analytical protocol):

* Compare outcomes in emergent stenting vs no stenting groups depending on stent subtype and endovascular approach
* Compare outcomes in emergent stenting vs no stenting groups depending on antithrombotic treatment before, during and after the endovascular procedure
* Define the potential impact of early statin treatment on the interplay between stenting vs no stenting and the outcomes.

STATISTICS:

Medians with IQRs and means with SDs together with percentages will be used to present the distribution of ordinal, continuous, and categorical variables. Baseline characteristics across groups will be compared using the Pearson χ2 test for categorical variables and t test or the Kruskal-Wallis test, as appropriate, for continuous and ordinal variables.

Given the nature of data deriving from prospective registries, inverse probability of treatment weighting (IPTW) will be implemented, which is an application of propensity scores that calculates the probability of being exposed to one treatment versus the other and creates a pseudo-population based on the probabilities so that potential confounders are equally distributed across the treatment groups.

Models will be weighted for prespecified variables known to potentially impact the outcome, and will also consider factors of imbalance between groups. In case of crossovers, a stratum-based analysis according to predefined estimand will be applied (direct intervention effect on outcomes and total-effect; estimand approach in detailed description).

DISSEMINATION The results will be disseminated in international peer reviewed journals.

CERES-TANDEM is promoted by

* Bufalini Stroke Center, AUSL Romagna, Cesena, Italy (PI Dr. M. Romoli)
* Interventional Neuroradiology Unit, Vall d'Hebron Institut de Recerca, Barcelona, Spain (PI Dr. F. Diana)
* Boston Medical Center and Boston University School of Medicine, Boston, Massachusetts, USA (PI Dr. T. Nguyen)

DETAILED DESCRIPTION:
BACKGROUND:

Tandem occlusion stroke, defined by concurrent extracranial and intracranial vessel occlusions, remains an underinvestigated subset of acute ischemic stroke. There is a critical gap in knowledge and data regarding tandem occlusion-related stroke treatment, mainly related to the very low inclusion rate of tandem stroke in endovascular thrombectomy trials, possibly in relation to the more severe features of tandem occlusion stroke.

The HERMES meta-analysis only had 122 participants with tandem occlusions, preventing from any inference on treatment effect and leading to a critical gap in current management guidelines (ESO-ESMINT guideline on mechanical thrombectomy 2019; TUrc et al., 2019).

While observational studies suggest potential benefits of emergent carotid stenting (eCAS), they also highlight risks such as hemorrhagic transformation and clinical deterioration, underscoring the need for large-scale data. Identification of features that could stratify the potential benefit of eCAS in patients with anterior circulation tandem occlusions could guide more individualised treatment strategies.

CERES-TANDEM is a multicenter study designed to improve the understanding of tandem ischemic stroke, with particular regard to the impact of emergent carotid stenting, early antithrombotic treatment, and early bleeding.

Objectives

Identify stroke risk factors: The prevalence and adjusted associations of traditional vascular risk factors-hypertension, diabetes mellitus, hypercholesterolaemia, smoking status, atrial fibrillation, prior stroke or transient ischaemic attack (TIA), and pre-stroke modified Rankin Scale (mRS)-between patients presenting with tandem cervical-intracranial occlusions and those with isolated large-vessel occlusions will be compared. Multivariable logistic regression will estimate odds ratios (ORs) for tandem versus single-site occlusion, adjusting for relevant covariates (age, sex).

Compare clinical outcomes of reperfusionIn both tandem-occlusion and isolated-occlusion cohorts, evaluating whether acute reperfusion therapies-intravenous thrombolysis, mechanical thrombectomy, and emergent carotid stenting-are associated with improved 3-month functional outcome. The estimate of the effect of each intervention versus medical management alone will be calculated using an inverse-probability-of-treatment-weighted (IPTW) ordinal logistic regression for shift in the full mRS distribution, and IPTW logistic regression for the dichotomous "good outcome" endpoint (mRS 0-2). Additional outcomes will adjust for baseline NIHSS, ASPECTS, onset-to-groin times, age and gender, and atrial fibrillation.

Assess post-stent therapy. Among patients undergoing emergent carotid stenting, a comparison of three post-procedural antithrombotic regimens-single antiplatelet, dual antiplatelet, and anticoagulation-on functional outcome, symptomatic intracranial haemorrhage (ECASS II definition), and recurrent ischaemic events within 90 days. IPTW-weighted logistic regression for binary endpoints will be used, with regimen as the exposure and adjustment for stent type, procedural variables, and baseline risk factors.

Study Design: A multicentre, observational cohort study pooling data from prospective stroke registries.

Inclusion criteria: adults (≥18 years) with acute ischaemic stroke due to anterior-circulation large-vessel occlusion treated between January 2018 and December 2024. Tandem occlusion defined as simultaneous extracranial internal carotid and intracranial large-vessel occlusion on imaging. Ethics approval was obtained at each site if needed; all data were de-identified under encrypted study IDs.

Data Collection: a predefined form available on solid support for offline use (constrined field dataset) and a RedCap CRFs will be available for data entry:

* Baseline variables (e.g. demographics, vascular risk factors, pre-stroke mRS, NIHSS on admission, onset-to-imaging time, ASPECTS, occlusion site)
* Imaging data: CT/CT-perfusion parameters, angiographic findings (TICI scores)
* Procedural details: stent subtype, access route, thrombolysis use, thrombectomy device, stenting sequence (anterograde vs retrograde), procedural duration.
* Medications
* Outcomes of interest at follow-up visits. Data completeness and consistency were monitored centrally; missingness patterns will be evaluated and handled via multiple imputation (Rubin's rules for pooling).

Statistical analysis:

All analyses will employ IPTW to emulate a randomised comparison: propensity scores for each treatment comparison will be estimated by logistic regression incorporating prespecified confounders (demographics, baseline stroke severity, imaging features, centre, calendar time). Loveplots will be used to display balance.

Ordinal outcomes: weighted proportional-odds models yielding common odds ratios (cORs) with 95% CIs; model fit and proportionality tested via score tests.

Binary outcomes: weighted logistic regression producing ORs. Subgroup and interaction analyses using IPTW model will be conducted for: pre-specified for large/medium vessel occlusion, access route, intravenous thrombolysis, antithrombotic intensity, and sedation.

Estimands:

All analyses will be conducted in accordance with the estimand framework (ICH E9(R1)). The investigators define a total-effect estimand using treatment-policy strategy, a controlled direct-effect estimand adjusting for post-treatment recanalization and bleeding, and a principal-stratum estimand restricting the population to never-crossers. The primary outcome will be compared between eCAS strategy and a no-stenting strategy in patients with tandem-occlusion stroke.

The primary estimand (treatment-policy centred) aims at identifying the effect of eCAS on mRS regardless of other interventional outcomes (total effect). The population includes all participants, with the eCAS group represented by those undergoing eCAS and no-stenting group including all those with any conservative treatment, regardless of any later crossover from the latter to the former. Stabilized weights will be applied in a weighted ordinal regression for the primary outcome to estimate the total effect (weighted ordinal regression; estimand 1), with results reported as common odds ratio (cOR) with 95% confidence intervals (CI) for shift in lower mRS score with eCAS vs no-stenting group. Secondary outcomes included excellent and good functional outcome. Additional outcomes (sICH, successful recanalization, END) were also calculated.

The investigators predefined an interaction analysis for access route, approach, large/medium vessel occlusion, type of sedation, IVT and periprocedural antithrombotic treatment intensity in the context of estimand 1, fitting a cumulative proportional regression and adjusting for age, sex, pre-stroke mRS, NIHSS at admission, ASPECTS, atrial fibrillation and OTG.

For estimand 1, the investigators prespecify a sensitivity analysis to account for the potential impact of successful intracranial recanalization on eCAS indication (reverse temporal association; sensitivity analysis on estimand 1).

A second estimand to identify the effect of eCAS on mRS not mediated by successful reperfusion or sICH (direct effect, estimand 2) will also be implemented. In the full cohort, successful recanalization (TICI 2b-3) and sICH were included as factors in the IPTW-weighted ordinal regression, reporting the adjusted cORs for eCAS (estimand 2).

A third principal-stratum estimand was planned, restricting the no-stenting group to participants who did not receive any treatment on the extracranial segment (excluding cases undergoing eCAS or any angioplasty procedure at the cervical occlusion site at the time of EVT or within 24 hours from EVT (estimand 3).

THe investigators will use R v4.3 for all analysis.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke
* tandem or isolated cervical artery occlusion (exploratory group)
* emergent extracranial vessel stenting or no stenting (treatment grouping variable)

Exclusion Criteria:

* hemorrhagic stroke
* no tandem occlusion and no isolated extracranial cervical vessel occlusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stroke due to tandem occlusion in the anterior or posterior circulation, and patients with stroke due to isolated cervical artery occlusion, independently from previous thrombolysis, antiplatelet or anticoagulant use
Sampling Method: Non-Probability Sample
Enrollment: 2880 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | 3 months
  modified Rankin Scale ranges 0 to 6, with 0 being optimal outcome (full autonomy) and 6 being mortality.

SECONDARY OUTCOMES:
symptomatic ICH | within the first 24 hours and within the first 7 days after stroke
  According to ECASS II criteria: any intracranial haemorrhage on any post-treatment image, within seven days of initiating treatment associated with a ≥ four-point deterioration on the NIHSS score from baseline or from the lowest score in seven days, or leading to death.
Any PH1-2 | within 7 days after intervention
  Any parenchymal hematoma 1-2
Early neurological deterioration | 48 hours
  4 or more points negative change in National Institutes of Health Stroke Scale (NIHSS, ranging 0 to 42, with 42 being tetraplegia and coma and 0 being no symptoms) within 24-48 hours from stroke. This will then be used in sub-strata according to etiology (hemorrhagic, thrombotic, no recanalization, unexplained).
mortality | 3 months
  mortality
Complications | 7 days
  e.g. SAH, vessel perforation, dissection, local hematoma
Post-treatment stent occlusion | <24 hours, 24 hours to 7 days, after day 7 (or after discharge from hospital)
  post-treatment stent occlusion

CONTACTS AND LOCATIONS:
Locations (3):
- Boston Medical Center, Boston, Massachusetts, United States
- Bufalini Hospital Comprehensive Stroke Center, Cesena, Italy
- Vall d'Hebron Institut de Recerca, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
to comply with privacy regulations (including GDPR)

REFERENCES:
- [Background] Diana F, Abdalkader M, Behme D, Li W, Maurer CJ, Pop R, Hwang YH, Bartolini B, Da Ros V, Bracco S, Cirillo L, Marnat G, Katsanos AH, Kaesmacher J, Fischer U, Aguiar de Sousa D, Peschillo S, Zini A, Tomasello A, Ribo M, Nguyen TN, Romoli M; APT-eCAS collaboration. Antithrombotic regimen in emergent carotid stenting for acute ischemic stroke due to tandem occlusion: a meta-analysis of aggregate data. J Neurointerv Surg. 2024 Feb 12;16(3):243-247. doi: 10.1136/jnis-2023-020204. PMID 37185107
- [Background] Diana F, Romoli M, Toccaceli G, Rouchaud A, Mounayer C, Romano DG, Di Salle F, Missori P, Zini A, Aguiar de Sousa D, Peschillo S. Emergent carotid stenting versus no stenting for acute ischemic stroke due to tandem occlusion: a meta-analysis. J Neurointerv Surg. 2023 May;15(5):428-432. doi: 10.1136/neurintsurg-2022-018683. Epub 2022 Apr 15. PMID 35428740
- [Derived] Romoli M, Molina CA, Zapata-Arriaza E, Jaikumar V, Jesser J, Heldner MR, Merlino G, Arba F, Giammello F, Radu RA, D'Anna L, Bigliardi G, Hanning U, Scarcia L, Puetz V, Abu Amara A, Zini A, Michel P, Aguiar De Sousa D, Al Kasab S, Casolla B, Kuhne Escola J, Da Ros V, Pezzini A, Candelaresi P, Alexandre AM, Toni D, Marto JP, Gabrieli JD, Sousa JA, Schwab R, Alpay K, Paciaroni M, Rapillo CM, Yeo L, Greisenegger S, Nolte CH, Caproni S, Anastasiou A, Tassi R, Maus V, Lattanzi S, Thanki SS, Sanna A, Naccarato M, Hawkes C, Abraham MG, Tudisco V, Requena M, Klein P, Ruggiero M, Lafe E, Medina-Rodriguez M, Monteiro A, Reiff T, Ringleb PA, Mohlenbruch M, Mujanovic A, Kaesmacher J, Peycheva M, Valente M, Taglialatela A, Toraldo F, Ferretti S, Toscano A, Ferrau L, Maffei S, Rosafio F, Schulte K, Kaiser D, Migliaccio L, Thevoz G, Soares MD, Abu Qdais A, Gardin A, Kohrmann M, Bellini L, Spina E, Andreone V, Nicolini E, Giacomozzi S, Sepe FN, Rosterman L, Aust A, Psychogios M, Selseth MN, Abdalkader M, Costalat V, Katsanos AH, Siddiqui AH, Longoni M, Tomasello A, Kristoffersen ES, Nguyen TN, Diana F; for CERES-TANDEM. Emergent Carotid Stenting for Acute Anterior Circulation Ischemic Stroke With Tandem Lesions: The Multicenter CERES-TANDEM Study. Neurology. 2026 Jan 27;106(2):e214528. doi: 10.1212/WNL.0000000000214528. Epub 2025 Dec 26. PMID 41453121